CLINICAL TRIAL: NCT05823246
Title: A Phase II Study to Evaluate the Efficacy and Safety of QLF31907 Injection in Patients With Advanced Melanoma and Urothelial Carcinoma
Brief Title: Safety and Efficacy Study of QLF31907 in Advanced Melanoma and Urothelial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QLF31907-201
Record Dates: First submitted 2023-03-10; First posted 2023-04-21 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-04

CONDITIONS: Melanoma; Urothelial Carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLF31907 (Experimental): single arm with QLF31907
  Interventions: Drug: QLF31907

INTERVENTIONS:
Drug: QLF31907 — Intravenous infusion once every two weeks. The dose administered in part 2 will depend on the outcome of part 1.

SUMMARY:
This study will assess the safety, tolerability and efficacy of every-2-week dosing of QLF31907 injection in patients with advanced melanoma and urothelial carcinoma.

DETAILED DESCRIPTION:
This study is divided into two parts. The first part is the safety and tolerability observation period, mainly observing the safety and tolerability of QLF31907. The second part is mainly the efficacy observation period, further evaluating the efficacy and safety of QLF31907 in patients with advanced melanoma and urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participated and signed a written informed consent form
2. Age ≥ 18 years, male or female
3. ECOG performance status of 0 or 1
4. Expected life-expectancy ≥ 3 months
5. Histologically confirmed diagnosis of locally advanced or metastatic unresectable melanoma or urothelial carcinoma, failed or intolerant or rejected to standard therapy
6. Patients must have at least one measurable lesion according to RECIST v1.1
7. Adequate organ function prior to QLF31907 administration
8. All subjects of reproductive potential must agree to use an effective method of contraception during the study and for 180 days after the last dose, and women of reproductive age must have a negative blood pregnancy result within 7 days prior to the first dose.

Exclusion Criteria:

1. Prior treatment with 4-1BB agonist or 4-1BB recombinant fusion protein
2. Known to be allergic to any excipients of QLF31907 or a history of severe allergic reactions to other monoclonal antibodies
3. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation, or autologous stem cell transplantation within 180 days
4. Known history of cytotherapy or antitumor vaccine or other antitumor therapy or surgical treatment of main organs within 4 weeks
5. Known history of systemic glucocorticoid therapy or other immunosuppressants within 14 days
6. Active central nervous system (CNS) metastases
7. Known history of other active malignant tumor within 3 years, unless completely cured
8. With uncontrolled or clinically symptomatic pleural, pericardial or abdominal effusions
9. An active infectious disease requiring intravenous antibiotic therapy
10. Failure to recover to grade 1 from adverse reactions due to prior treatment according to CTCAE v5.0
11. An active autoimmune diseases or known history of ≥ grade 3 irAE due to prior immunotherapy
12. Known history of active hepatitis B/C infection, severe cardiovascular and cerebrovascular disease, idiopathic pulmonary fibrosis, pneumoconiosis, asbestosis, hepatitis (nonalcoholic steatohepatitis, alcoholic or autoimmune hepatitis), cirrhosis, active tuberculosis, active syphilis, HIV infection
13. Poorly controlled respiratory, circulatory or endocrine diseases
14. Known history of drugs abuse, alcoholism, neurologic or psychiatric disorders
15. Patients who are breastfeeding
16. Other serious physical or psychiatric illnesses or laboratory abnormalities that may increase the risk of participating in the study, or interfere with the results of the study, and patients who are not suitable for participation in this study in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
(part 1)Dose-limiting toxicity(DLT) | 28days
(part 2) Objective response rate(ORR) | up to 2 years

SECONDARY OUTCOMES:
(part 2) Safety index: adverse event(AE), serious adverse event (SAE), treatment-related adverse event(TRAE) | up to 2 years
(part 2) Progression-free survival(PFS) | up to 2 years
(part 2) Overall survival(OS) | up to 2 years
(part 2) Maximum observed plasma concentration (Cmax) | up to 2 years
(part 2) Positive rate of anti-drug antibody(ADA) | up to 2 years

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - West China Hospital, Chengdu, Sichuan